CLINICAL TRIAL: NCT00940472
Title: Randomized, Double-Blind, Efficacy and Safety, Controlled Study, Between DMMET-01 and Metformin on Improvement of Metabolic Control in Naive Type 2 Diabetics Patients.
Brief Title: Study on DMMET-01 Versus Metformin on Improvement of Metabolic Control in Naive Type 2 Diabetes Patients
Acronym: DMMET2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Jorge González Canudas/Medical director, Silanes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-0790/2009; SIL-DMMET080609
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Diabetes Type 2
Keywords: type 2 diabetes; monotherapy; antidiabetics; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Drug (Experimental): DMMET-01 + Diet
  Interventions: Drug: DMMET-01
- Metformin (Active Comparator): Metformin + Diet
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: DMMET-01 — 90 days: 15 days daily dose 1050.6 mg (before dinner)+75 days dose twice a day 1050.6 mg (before breakfast) 1050.6 mg (before dinner).
  Arms: Experimental Drug
Drug: Metformin Hydrochloride — 90 days: 15 days daily dose 850 mg (before dinner)+ 75 days dose twice a day 850 mg (before breakfast) 850 mg (before dinner)
  Other Names: Comparator
  Arms: Metformin

SUMMARY:
The aim of this clinical trial is to compare the efficacy of DMMET-01 versus metformin hydrocloride on metabolic control in mexican type 2 diabetes patients without prior pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study: 40 to 60 years
* With type 2 diabetes evolution < 5 years without pharmacological treatment 1 month prior to the screening
* Fasting glucose = 130-200 mg/dL
* HbA1c of 7% to 9%
* Blood pressure < 140/80 mmHg
* Ability to communicate and meet the requirements of the study
* Signed Written Informed Consent before to conducting any study
* Body mass index (BMI) of 25 kg/m2 to 35 Kg/m2

Exclusion Criteria:

* Suspected or confirmed pregnancy
* Nursing
* Inability to secure the non-pregnant during the study duration
* Hypersensitivity to any biguanides
* Use of an investigational drug within 30 days prior to the screening
* Liver failure, heart failure, kidney failure or thyroid disease
* Periods of acute or chronic diarrhea or vomiting
* Chronic hepatic disease
* Total Cholesterol >300 mg/dL
* Triglycerides >400 mg/dL

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Metabolic Control (Fasting glucose, postprandial glucose, HbA1C) | 3 months

SECONDARY OUTCOMES:
Lipid Profile (Total cholesterol, HDL, LDL, triglycerides) | 3 months
Adverse Events | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A González, MD, Study Director — Laboratorios Silanes S.A. de C.V.; Manuel González, PHD, Study Chair — University of Guadalajara; Esperanza Martínez, PHD, Principal Investigator — University of Guadalajara
Locations (1):
- Centro Universitario de Ciencias de la Salud, Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Aguilar-Salinas CA, Velazquez Monroy O, Gomez-Perez FJ, Gonzalez Chavez A, Esqueda AL, Molina Cuevas V, Rull-Rodrigo JA, Tapia Conyer R; Encuesta Nacional de Salud 2000 Group. Characteristics of patients with type 2 diabetes in Mexico: Results from a large population-based nationwide survey. Diabetes Care. 2003 Jul;26(7):2021-6. doi: 10.2337/diacare.26.7.2021. PMID 12832306
- [Background] González-Ortiz M, Martínez-Abundis E. Síndrome de resistencia a la insulina. En, Diabetes mellitus. Islas-Andrade S, Revilla-Monsalve C. McGrawHill-Interamericana. 3a. edición. México, 2005. ISBN p. 203-14.
- [Background] Gonzalez-Ortiz M, Martinez-Abundis E, Kam-Ramos AM, Hernandez-Salazar E, Ramos-Zavala MG. Effect of ezetimibe on insulin sensitivity and lipid profile in obese and dyslipidaemic patients. Cardiovasc Drugs Ther. 2006 Apr;20(2):143-6. doi: 10.1007/s10557-006-7805-x. PMID 16761194
- [Background] Gonzalez-Ortiz M, Martinez-Abundis E; Grupo para el Tratamiento de la Diabetes Mellitus con Combinaciones. [Efficacy and safety of glimepiride plus metformin in a single presentation, as combined therapy, in patients with type 2 diabetes mellitus and secondary failure to glibenclamide, as monotherapy]. Rev Invest Clin. 2004 May-Jun;56(3):327-33. Spanish. PMID 15612515
- [Background] American Diabetes Association. Standards of medical care in diabetes--2007. Diabetes Care. 2007 Jan;30 Suppl 1:S4-S41. doi: 10.2337/dc07-S004. No abstract available. PMID 17192377
- [Background] Jeyaseelan L, Rao PS. Methods of determining sample sizes in clinical trials. Indian Pediatr. 1989 Feb;26(2):115-21. PMID 2753525